CLINICAL TRIAL: NCT02020629
Title: Effect of Lixisenatide on Glucagon Secretion During Hypoglycemia in Patients With Insulin-treated Type 2 Diabetes
Brief Title: Study on Lixisenatide and Counterregulation to Hypoglycemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Bo Ahren, Professor, Lund University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16; 2012-004959-36 (EudraCT Number)
Record Dates: First submitted 2013-12-16; First posted 2013-12-25 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Type 2 Diabetes
Keywords: Glucagon; Hypoglycemia; Counterregulation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia | interventions — lixisenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lixisenatide (Experimental): Lixisenatide 20µg daily
  Interventions: Drug: Lixisenatide

INTERVENTIONS:
Drug: Lixisenatide — Lixisenatide is given for 6 weeks whereafter a hypoglycemia clamp is undertaken
  Other Names: Lyxumia

SUMMARY:
In hypoglycemia, there is a counterregulation to restore glucose levels. An important part of this counterregulation is the release of the hormone glucagon. Since the GLP-1 receptor agonist lixisenatide has been shown to be associated with a low risk of hypoglycemia, this study examines whether lixisenatide affects the glucagon response to hypoglycemia.

DETAILED DESCRIPTION:
The study is a single-center, randomized, placebo-controlled study with a cross-over design and examines the glucagon response during a hyperinsulinemic hypoglycemic phase after a 6-week treatment with lixisenatide (or placebo) as add-on to basal insulin and metformin. The hypothesis of the study is that the glucagon counterregulation to hypoglycemia in patients treated with lixisenatide and basal insulin is not lower than in patients treated with basal insulin.

ELIGIBILITY:
Inclusion Criteria:

1. Male, non-fertile female or female of childbearing potential using a medically approved birth control method aged >18 years.
2. Adult patients with type 2 diabetes treated with basal insulin (NPH insulin, insulin detemir, insulin glargine or insulin degludec) (stable insulin dose (±10%) during the last three months) with concomitant at >3 months stable dose (>1500 mg daily) of metformin.
3. HbA1c <10% (DCCT standard; < 83 mmol(mol) at visit 1.

Exclusion Criteria:

1. Treatment with antihyperglycemic agents apart from basal insulin and metformin, i.e., bolus insulin or other antihyperglycemic oral agents apart from metformin
2. Type 1 diabetes (including LADA)
3. Pregnant or lactating female. Women of childbearing potential with no effective contraceptive method. Acceptable contraceptive include contraceptive sponge; hormonal contraception pills, patches, vaginal rings, injectable contraceptives; and intrauterine devices. Women of childbearing potential (pre-menopausal, not surgically sterile women for at least 3 months prior to the time of screening) must have a confirmed negative serum pregnancy test at screening visit. They must use an effective contraceptive method throughout the study, and agree to repeat pregnancy tests at designated visits. The applied methods of contraception have to meet the criteria for a highly effective method of birth control according to the "Note for guidance on non-clinical safety studies for the conduct of human clinical trials for pharmaceuticals (CPMP/ICH/286/95)"
4. A history of any secondary forms of diabetes, e.g., Cushing's syndrome and acromegaly.
5. Acute infections which may affect blood glucose control within 4 weeks prior to visit 1
6. Any history of recent (<2 weeks) recurrent or severe hypoglycemic episodes or hypoglycemia unawareness
7. Donation of one unit (500 ml) or more of blood, significant blood loss equaling to at least one unit of blood within the past 2 weeks or a blood transfusion within the past 8 weeks.
8. Treatment with growth hormone and oral or parenteral corticosteroid (> 7 consecutive days of treatment) within 8 weeks prior to visit 1 and thereafter during the whole study period.
9. Use of other investigational drugs within 30 days prior to visit 1.
10. Laboratory findings at the time of screening, including amylase and/or lipase > 3 times the upper limit of the normal laboratory range (ULN) and P-calcitonin ≥20 pg/ml (5.9 pmol/L).
11. Personal or immediate family history of medullary thyroid cancer (MTC) or genetic condition that predisposes to MTC (e.g. multiple endocrine neoplasia syndromes).
12. History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery
13. Allergic reaction to any GLP-1 receptor agonist or to metacresol
14. Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting,
15. Cardiovascular, hepatic, neurological, or endocrine disease, active malignant tumor or other major systemic disease or patients with short life expectancy making implementation of the protocol or interpretation of the study results difficult.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Glucagon response to hypoglycemia | 30 min
  Hypoglycemia is induced by clamp during 30 min; glucagon levels are measured during this time frame

SECONDARY OUTCOMES:
Cortisol response to hypoglycemia | 30 min
  Hypoglycemia is induced by a clamp during 30 min. Cortisol is measured during this time frame.
Catecholamines | 30 min
  Hypoglycemia is induced by a clamp during 30 min. Catecholamines are measured during this time frame.

OTHER OUTCOMES:
HbA1c | 6 weeks
  Change in HbA1c during six weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bo Ahrén, MD, PhD, Principal Investigator — Lund University
Locations (1):
- Clinical Research Department, Malmo, Sweden

REFERENCES:
- [Derived] Farngren J, Persson M, Ahren B. Effect of the GLP-1 Receptor Agonist Lixisenatide on Counterregulatory Responses to Hypoglycemia in Subjects With Insulin-Treated Type 2 Diabetes. Diabetes Care. 2016 Feb;39(2):242-9. doi: 10.2337/dc15-1274. Epub 2015 Nov 4. PMID 26537183